CLINICAL TRIAL: NCT05233163
Title: Sodium-Glucose Cotransporter-2 (SGLT2) Inhibitors in Transthyretin Amyloid (ATTR) Cardiomyopathy
Brief Title: SGLT2 Inhibitors in Transthyretin Amyloid Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mathew S. Maurer, MD, Arnold and Arlene Goldstein Professor of Cardiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT9709
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Transthyretin Amyloid Cardiomyopathy
Keywords: Sodium-glucose cotransporter 2 inhibitor (SGLT2i); Empagliflozin; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Drug Arm (Experimental): Subjects will take empagliflozin 10 mg oral daily for 12 weeks.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10 mg oral daily for 12 weeks
  Other Names: Jardiance

SUMMARY:
This is a single center, single arm, prospective, 12 week open label pilot trial of the sodium-glucose cotransporter 2 inhibitor (SGLT2i), empagliflozin 10 mg oral daily, in patients with transthyretin amyloid cardiomyopathy (ATTR-CM). The target population for enrollment will be subjects with ATTR-CM and either non-insulin dependent diabetes mellitus or chronic kidney disease. The primary aim will be to assess the safety and tolerability of empagliflozin 10 mg oral daily in subjects with heart failure secondary to ATTR, which remain unexplored. The accrual target is 15 subjects. Consented subjects will be evaluated for safety and tolerability of study drug, empagliflozin 10 mg oral daily, over a period of 12 weeks. Subjects will undergo a total of 6 study visits: 3 in-person and 3 telephone follow-ups.

DETAILED DESCRIPTION:
Transthyretin amyloid cardiomyopathy (ATTR-CM) is an underrecognized cause of heart failure among older adults, in which misfolded transthyretin (TTR) proteins build up in the muscle tissue of the heart. In 2018, a drug called tafamidis was proven to stabilize the protein and protect people from further damage, and in 2019, it was approved for use in ATTR-CM by the U.S. Food and Drug Administration (FDA). But while people with ATTR-CM are living longer, they continue to suffer from symptoms of heart failure and cardiorenal syndrome as the disease progresses. Sodium glucose co-transporter inhibitors (SGLT2i) are drugs used to treat diabetes mellitus, heart failure, and chronic kidney disease. They may also reduce systemic inflammation, and affect body composition (fat, lean mass, and total water contents) in patients with heart failure, a condition which also has significant overlap with obesity. No one has explored the safety, tolerability, and clinical effects of SGLT2i in patients with heart failure due to ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

* Every participant must meet all of the following inclusion criteria to be eligible for enrollment in this study:

  1. Age ≥ 18 years old
  2. Diagnosis of TTR cardiac amyloidosis (wild type or variant), confirmed by the presence of amyloid deposits on analysis of biopsy specimens obtained from cardiac and noncardiac sites (e.g. fat aspirate, gastrointestinal sites, salivary glands, or bone marrow), technetium-99m pyrophosphate cardiac scintigraphy, or mass spectrometry
  3. Normal serum free light chain ratio and the absence of abnormal monoclonal band on serum and urine immunofixation
  4. Subjects will have at least 1 of the indications below for an SGLT2i, and meet package-insert criteria for drug initiation: non-insulin dependent diabetes mellitus with hemoglobin A1c ranging from 6.5-9.9 OR chronic kidney disease (defined as an estimated glomerular filtration rate of 25-75 ml/minute/1.73 m2 of body-surface area)
  5. On stable oral diuretics (defined as no more than a 50% increase from baseline diuretic dose established during a sustained 2 week period) within 2 weeks before enrollment
  6. Able to understand and sign the informed consent document after the nature of the study has been fully explained

Exclusion Criteria:

* The presence of any of the following excludes eligibility for enrollment in this study:

  1. Prior liver or heart transplantation
  2. Active malignancy or non-amyloid disease with expected survival of less than 1 year
  3. Heart failure, in the opinion of the investigator, primarily caused by severe left-sided valve disease. Note: if valve was repaired, subject may be considered as no longer with severe valve disease
  4. Heart failure, in the opinion of the investigator, primarily caused by ischemic heart disease
  5. Ventricular assist device or anticipated within the next 6 months
  6. Pacemaker or implantable cardioverter defibrillator incompatible with magnetic resonance technology
  7. Absolute contraindication for quantitative magnetic resonance (e.g. aneurysmal clips, metal objects)
  8. Impairment from stroke, injury or other medical disorder that precludes participation in the study
  9. Myocardial infarction, cardiovascular surgery, stroke or transient ischemic attack within the prior 90 days
  10. Disabling dementia or other mental or behavioral disease
  11. Enrollment in a clinical trial not approved for co-enrollment
  12. Expected use of continuous intravenous inotropic therapy in the next 6 months
  13. High risk for non-adherence as determined by screening evaluation
  14. Inability or unwillingness to comply with the study requirements
  15. Chronic kidney disease with estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2 or end-stage renal disease
  16. Current or prior SGLT2i use
  17. Type 1 diabetes mellitus or insulin-dependent diabetes mellitus
  18. N-terminal (NT)-pro hormone BNP (NT-proBNP) < 300 pg/mL or < 900 pg/mL if concomitant diagnosis of atrial fibrillation
  19. History of ketoacidosis
  20. History of complex urinary tract or genital infections
  21. History of kidney stone
  22. Systolic blood pressure < 90 mmHg and symptomatic hypotension
  23. Systolic blood pressure ≥ 180 mmg Hg
  24. Chronic obstructive pulmonary disease
  25. Major surgery in the 90 days before or after screening
  26. Chronic alcohol or drug abuse
  27. Nursing home resident
  28. Other reason that would make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Maurer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin: Participants will take empagliflozin 10 mg oral daily for 12 weeks.
Period: Overall Study
Arm/Group | Empagliflozin
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 81 [72 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
Participants | 0

2. Secondary Outcome: Mean Change in Daily Diuretic Dose
Description: Calculated in mg/kg of furosemide equivalence. This outcome was assessed at Baseline, 6 weeks, and 12 weeks; the change from baseline to 12 weeks is reported.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
mg/kg | -12 [-21 to -3]

3. Secondary Outcome: Mean Change in Body Weight
Description: Change in body weight (kg) at trial end compared to trial start
Time Frame: Baseline, 6 weeks and 12 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
kg | -0.97 [-1.73 to -0.21]

4. Secondary Outcome: Mean Change in Total Water Content
Description: Change in total water content (kg) as assessed by bioimpedance analysis and quantitative magnetic resonance techniques at trial end compared to trial start
Time Frame: Baseline, 6 weeks and 12 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
kg | -0.63 [-1.22 to -0.04]

5. Secondary Outcome: Mean Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent (better outcome). This outcome was assessed at Baseline, 6 weeks, and 12 weeks; the change from baseline to 12 weeks is reported.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
score on a scale | 4 [-2 to 10]

6. Secondary Outcome: Mean Change in Short Physical Performance Battery Score
Description: The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons. Each test is scored on a 0 to 4 scale using previously validated norms and summed for an overall score range of 0 to 12, with 0 indicating the lowest physical performance, and scores of 12 indicating the highest performance (better outcome). This outcome was assessed at Baseline, 6 weeks, and 12 weeks; the change from baseline to 12 weeks is reported.
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Empagliflozin
Number analyzed (Participants) | 15
score on a scale | -0.7 [-2 to 1]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Empagliflozin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin (N=15)
Transient episode of symptomatic hypotension (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Increased urination (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Eye stye (Eye disorders) | 1
Symptomatic COVID-19 (Infections and infestations) | 3
Headache (General disorders) | 1
Leg cramping (General disorders) | 1
Lower extremity pruritus (General disorders) | 1
Sinusitis (General disorders) | 1
Lower extremity wound infection (Infections and infestations) | 1 — Skin trauma prior to study enrollment; initial improvement followed by subsequent worsening of wound
Floaters (Eye disorders) | 1
Mechanical fall (Injury, poisoning and procedural complications) | 2
Tingling sensation in arm (General disorders) | 1
Foot pain, acute onset (General disorders) | 1
Head congestion (General disorders) | 2
Muscle pain (Musculoskeletal and connective tissue disorders) | 3
Irregular heart rate (Cardiac disorders) | 1
Disruption in taste and appetite (General disorders) | 1
Bilateral groin intertrigo (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT05233163/Prot_SAP_000.pdf